CLINICAL TRIAL: NCT05992558
Title: Development of Longitudinal Multimarker Risk Models for Decision Support Across the Clinical Follow-up of Very Elderly Patients With Heart Failure and Preserved Ejection Fraction
Brief Title: Longitudinal Multimarker Risk Models for Very Elderly Patients With Heart Failure and Preserved Ejection Fraction
Status: Active, not recruiting | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); European Union (Other)
Responsible Party: Sponsor
Other Study IDs: PI21/00541
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Preserved Ejection Fraction; Elderly; Prognostic model; Risk; Hospitalization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Serum, EDTA plasma, lithium heparin plasma, and buffy coat.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Very elderly HFpEF: Prospective cohort of very elderly patients (≥80 years old) with heart failure with preserved ejection fraction (HFpEF) consecutively admitted for acute HF

SUMMARY:
The goal of this observational study is to develop longitudinal multimarker risk models for decision support during the clinical follow-up of very elderly patients with heart failure and preserved ejection fraction (HFpEF).

The main questions it aims to answer are:

* Can advanced risk prediction models accurately estimate the prognosis of very elderly patients with HFpEF over a 1-year follow-up after a hospitalization for acute heart failure?
* Do novel biomarkers, in addition to routine clinical variables and elderly-specific predictors, contribute to improved risk prediction for these patients?

To this end, very elderly patients (aged 80 or older) who have HFpEF and were admitted for acute heart failure will be included. Clinical and biological data will be collected during their hospitalization and also during follow-up visits 30 and 90 days after discharge.

There is no comparison group in this observational study.

DETAILED DESCRIPTION:
Background: Very elderly patients with heart failure and preserved ejection fraction (HFpEF) are under-represented in risk prediction models, and the role of prognostic biomarkers in this population is unclear due to the presence of cumulative comorbidity burden. Risk prediction is a useful tool to support decision making across the clinical follow-up of very elderly HFpEF patients.

Aim: To develop longitudinal prognostic models based on readily available clinical and biological variables, novel biomarkers and elderly-specific predictors to estimate prognosis over 1-year follow-up after a HF hospitalization in very elderly patients with HFpEF.

Design: Observational, single-centre, prospective cohort study of very elderly patients (≥80 years old) with HFpEF consecutively admitted for acute HF.

Main outcome: Composite of 1-year all-cause mortality and/or HF-hospitalization. Sample size: 184 patients.

Follow-up time: 1 year. Predictors: Routine clinical variables (sociodemographic, medical history, physical examination, vital signs, laboratory tests, imaging, concomitant medication, quality of life and elderly-specific factors) and novel biomarkers will be longitudinally collected during index hospitalization, 30-day and 90-day post-discharge visits.

Statistical analysis: Kaplan-meier survival analysis. Logistic and Cox proportional-hazards regression models, time-to-event models for repeated events, linear-mixed effects, joint models, LASSO and machine learning techniques will be used for model development.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥80 years;
2. diagnosis of HFpEF, requiring the 4 following conditions: b1) typical symptoms and/or signs of HF; b2) left ventricular ejection fraction (LVEF) ≥50%; b3) elevated levels of natriuretic peptides (NTproBNP ≥300 pg/mL or BNP ≥100 pg/mL in sinus rhythm; NT-proBNP ≥900 pg/mL or BNP ≥300 pg/mL in atrial fibrillation); and b4) at least one additional criterion: b4.1) relevant structural heart disease (left ventricular hypertrophy and/or left atrial enlargement), or 4.2) diastolic dysfunction;
3. hospitalization with a primary diagnosis of acute HF; and
4. giving informed consent.

Exclusion Criteria:

1. any clinical condition, such as HF secondary to congenital heart disease and severe valve disease, severe renal (requiring dialysis) and liver disease, active malignant diseases, autoimmune diseases, other diseases resulting in <1-year life expectancy or any other condition that, according to investigators' criteria, could significantly interfere with the study objectives;
2. any clinical or social condition that prevents clinical follow-up.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Very elderly patients (≥80 years old) with HFpEF consecutively admitted for acute HF at Hospital Universitario Ramón y Cajal and followed up at Unit of Heart Failure (UICA) of the Internal Medicine Dept.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Composite of 1-year all-cause mortality and/or HF-hospitalization | 12 months
  Combined outcome of all-cause mortality and/or readmission for acute heart failure during a 12-month follow-up period after index hospitalization

SECONDARY OUTCOMES:
1-year HF-hospitalization | 12 months
  Readmission for acute heart failure during a 12-month follow-up period after index hospitalization
3-month HF-hospitalization | 3 months
  Readmission for acute heart failure during a 3-month follow-up period after index hospitalization
1-month HF-hospitalization | 1 month
  Readmission for acute heart failure during a 1-month follow-up period after index hospitalization
1-year all-cause hospitalization | 12 months
  All-cause readmission during a 12-month follow-up period after index hospitalization
3-month all-cause hospitalization | 3 months
  All-cause readmission during a 3-month follow-up period after index hospitalization
1-month all-cause hospitalization | 1 month
  All-cause readmission during a 1-month follow-up period after index hospitalization
1-year all-cause mortality | 12 months
  All-cause mortality during a 12-month follow-up period after index hospitalization
1-year cardiovascular mortality | 12 months
  Cardiovascular mortality during a 12-month follow-up period after index hospitalization
1-year urgent HF visits | 12 months
  Urgent or unscheduled visit with new or worsening symptoms of acute heart failure requiring initiation of intravenous diuretic or vasoactive agent or mechanical or surgical intervention, with no hospital admission, during a 12-month follow-up period after index hospitalization
3-month urgent HF visits | 3 months
  Urgent or unscheduled visit with new or worsening symptoms of acute heart failure requiring initiation of intravenous diuretic or vasoactive agent or mechanical or surgical intervention, with no hospital admission, during a 3-month follow-up period after index hospitalization
1-month urgent HF visits | 1 month
  Urgent or unscheduled visit with new or worsening symptoms of acute heart failure requiring initiation of intravenous diuretic or vasoactive agent or mechanical or surgical intervention, with no hospital admission, during a 1-month follow-up period after index hospitalization
1-year worsening in NYHA class | 12 months
  Worsening of New York Heart Association (NYHA) Functional Classification (Class I to IV) at 12 months from the index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Manzano Espinosa, MD PhD, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
After the end of the project, the generated dataset and the metadata file will be deposited in an open data repository, complying with open science criteria - FAIR.
  Moreover, study documentation, including study protocol, statistical analysis and informed consent form will be shared openly.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From 1 year after the end of the project and for at least 5 years.
Access Criteria: IPD will be available to stakeholders, authorities, ethics committees and other parties legitimately interested in verifying their proper treatment and management.
  IPD may be used to ensure the scientific quality of the project results. That is to say, to carry out reproducibility of the results, if necessary at the request of scientific publication entities, among others, with prior authorization from the Research Ethics Committee, they may be reused for new research projects, provided that the consent collected allows it and/or in accordance with the applicable laws on data protection.

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):1757-1780. doi: 10.1016/j.jacc.2021.12.011. Epub 2022 Apr 1. PMID 35379504
- [Background] Taylor CJ, Moore J, O'Flynn N. Diagnosis and management of chronic heart failure: NICE guideline update 2018. Br J Gen Pract. 2019 May;69(682):265-266. doi: 10.3399/bjgp19X702665. No abstract available. PMID 31023695
- [Background] Sicras-Mainar A, Sicras-Navarro A, Palacios B, Varela L, Delgado JF. Epidemiology and treatment of heart failure in Spain: the HF-PATHWAYS study. Rev Esp Cardiol (Engl Ed). 2022 Jan;75(1):31-38. doi: 10.1016/j.rec.2020.09.033. Epub 2020 Dec 27. English, Spanish. PMID 33380382
- [Background] Kuster N, Huet F, Dupuy AM, Akodad M, Battistella P, Agullo A, Leclercq F, Kalmanovich E, Meilhac A, Aguilhon S, Cristol JP, Roubille F. Multimarker approach including CRP, sST2 and GDF-15 for prognostic stratification in stable heart failure. ESC Heart Fail. 2020 Oct;7(5):2230-2239. doi: 10.1002/ehf2.12680. Epub 2020 Jul 10. PMID 32649062
- [Background] Nunez J, Bayes-Genis A, Revuelta-Lopez E, Ter Maaten JM, Minana G, Barallat J, Cserkoova A, Bodi V, Fernandez-Cisnal A, Nunez E, Sanchis J, Lang C, Ng LL, Metra M, Voors AA. Clinical Role of CA125 in Worsening Heart Failure: A BIOSTAT-CHF Study Subanalysis. JACC Heart Fail. 2020 May;8(5):386-397. doi: 10.1016/j.jchf.2019.12.005. Epub 2020 Mar 11. PMID 32171764
- [Background] Pacho C, Domingo M, Nunez R, Lupon J, Nunez J, Barallat J, Moliner P, de Antonio M, Santesmases J, Cediel G, Roura S, Pastor MC, Tor J, Bayes-Genis A. Predictive biomarkers for death and rehospitalization in comorbid frail elderly heart failure patients. BMC Geriatr. 2018 May 9;18(1):109. doi: 10.1186/s12877-018-0807-2. PMID 29743019
- [Background] Levy WC, Mozaffarian D, Linker DT, Sutradhar SC, Anker SD, Cropp AB, Anand I, Maggioni A, Burton P, Sullivan MD, Pitt B, Poole-Wilson PA, Mann DL, Packer M. The Seattle Heart Failure Model: prediction of survival in heart failure. Circulation. 2006 Mar 21;113(11):1424-33. doi: 10.1161/CIRCULATIONAHA.105.584102. Epub 2006 Mar 13. PMID 16534009